CLINICAL TRIAL: NCT03504033
Title: Xenon-anesthesia on Patients Undergoing Major Liver-resection: Randomized Controlled Trial
Brief Title: Xenon-anesthesia on Patients Undergoing Major Liver-resection
Acronym: XeLiv
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: A device would have had to be maintained. The maintenance company is insolvent; both another maintenance company and another serviced device were not available.
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-163
Record Dates: First submitted 2018-03-14; First posted 2018-04-20 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Liver Function After Partial Liver Resection
Keywords: Xenon; Liver resection; post-operative liver failure; anesthetics, inhalation; Desflurane; Randomized controlled trail; RCT
MeSH Terms: conditions — Respiratory Aspiration | interventions — Xenon; Desflurane

STUDY DESIGN:
Intervention Model Description: Single-center, controlled, double-blinded, randomized, two-arm parallel, interventional clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This trial will be performed double-blinded. After randomization neither the patients nor the investigator of the baseline assessment and the postoperative assessment will be aware of the treatment allocation. The intraoperative anesthesiologist will not be blinded, due to feasibility and safety reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenon (Experimental): Xenon concentration of 50-60 % will be used for maintenance of general anesthesia and will be adjusted to maintain Bispectral index (BIS) value between 40 and 60.
  Interventions: Drug: Xenon
- Desflurane (Active Comparator): Desflurane concentrations of 4-5%/0.8 minimum alveolar concentration (MAC) respectively will be used for maintenance of general anesthesia and will be adjusted to maintain BIS index value between 40 and 60.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Xenon — inhalation to maintain anesthesia
  Other Names: LenoXe
  Arms: Xenon
Drug: Desflurane — inhalation to maintain anesthesia
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
The aim of this study is to compare the postoperative outcome of patients undergoing major liver resection under xenon- compared to desflurane-anesthesia.

DETAILED DESCRIPTION:
The aim of this study is to compare the postoperative liver function and additional outcome parameters of patients undergoing major liver resection under xenon- compared to desflurane-anesthesia. Xenon is known to maintain hemodynamic stability and consecutive tissue perfusion. Together with its potential for ischemic pre-conditioning, we hypothesize a protective effect of xenon on post-operative liver failure and ischemia/reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 3 segments liver resection
* ≥ 18 years
* Both gender
* American Society of Anesthesiologists (ASA) classification I-III
* Written informed consent prior to study participation

Exclusion Criteria:

Subjects, fulfilling one or more of the following exclusion criteria will not be included in the study:

* Severe pulmonary or airway disease
* Severe liver disease, accompanied by a Child-Pugh class >A
* Allergy/hypersensitivity to study medications
* ASA ≥ IV
* Patients susceptible to malignant hyperthermia
* Women who are pregnant, breast-feeding or women of childbearing potential not using adequate contraceptive methods
* Patients with preeclampsia or eclampsia
* Patients legally unable to give written informed consent.
* Patients with risk of high oxygen demand
* Patient with seriously impaired cardiac function
* All contraindications for xenon anesthesia according to the summary of product characteristics LENOXe
* Patient participates in a parallel interventional clinical trial during this study or receives an investigational drug within 30 days prior to inclusion into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-11 (Estimated); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Time-course of postoperative liver injury and function | Within the first 7 postoperative days
  The primary study outcome is the difference in postoperative liver injury and function between the two study arms, measured by the perioperative time-course of the liver transaminase alanine-aminotransferase (ALAT) preoperative and on postoperative days (POD) 1-3, 5 and 7.

SECONDARY OUTCOMES:
Intra- and postoperative blood loss | Surgery and ICU stay (maximum POD 7)
  Difference of intra- and postoperative blood loss between the two study arms until discharge from ICU or POD 7 (whichever occurs first)
Quantity of intra- and postoperative infusions | Surgery and ICU stay (maximum POD 7)
  Difference in quantity of infused crystalloids abd colloids between the two study arms until discharge from ICU or POD 7 (whichever occurs first)
Quantity of intra- and postoperative blood products | Surgery and ICU stay (maximum POD 7)
  Difference in quantity of transfused packed red blood cells (RBCs), fresh frozen plasma (FFP) and platelet concentrates between the two study arms until discharge from ICU or POD 7 (whichever occurs first)
Quantity of intra- and postoperative coagulation products | Surgery and ICU stay (maximum POD 7)
  Difference in quantity of administered tranexamic acid, fibrinogen and prothrombin complex concentrates between the two study arms until discharge from ICU or POD 7 (whichever occurs first)
Necessity and duration of surgical pringle maneuver | Surgery
  Difference in necessity and duration of intraoperative pringle maneuver performed by the surgeon between study groups
Necessity and duration of surgical total vascular occlusion | Surgery
  Difference in necessity and duration of intraoperative total vascular occlusion performed by the surgeon between study groups
Surgery time | Surgery
  Difference in surgery time between study groups
Fibrosis in the resected liver tissue | Surgery
  Difference in fibrosis in the resected liver tissue between the two study arms
Number of hepatocytes in synthesis phase in the resected liver tissue | Surgery
  Difference in number of hepatocytes in synthesis phase in the resected liver tissue between the two study arms
Number of macrophages in the resected liver tissue | Surgery
  Difference in number of macrophages in the resected liver tissue between the two study arms
Expression of Interleukin 6 (IL-6) in the resected liver tissue | Surgery
  Difference in expression of Interleukin 6 (IL-6) in the resected liver tissue between the two study arms
Expression of tumor necrosis factor (TNF) in the resected liver tissue | Surgery
  Difference in expression of tumor necrosis factor (TNF) in the resected liver tissue between the two study arms
Expression of hepatocyte growth factor (HGF) in the resected liver tissue | Surgery
  Difference in expression of hepatocyte growth factor (HGF) in the resected liver tissue between the two study arms
Expression of epidermal growth factor (EGF) in the resected liver tissue | Surgery
  Difference in expression of epidermal growth factor (EGF) in the resected liver tissue between the two study arms
Expression of fibroblast growth factor (FGF) in the resected liver tissue | Surgery
  Difference in expression of fibroblast growth factor (FGF) in the resected liver tissue between the two study arms
Expression of insulin-like growth factors I/II (IGF-I/II) in the resected liver tissue | Surgery
  Difference in expression of insulin-like growth factors I/II (IGF-I/II) in the resected liver tissue between the two study arms
Weight of the resected liver tissue | Surgery
  Difference in weight of the resected liver tissue normalized to body weight (%BW) between the two study arms
Computer tomography-assisted planimetry of the resected liver tissue | Surgery
  Difference in area of the resected liver tissue, assessed with computer tomography assisted planimetry, between the two study arms
Time-course of hemoglobin (Hb) | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of hemoglobin (Hb), between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of platelet count | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of platelet count, between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of prothrombin time (PT) | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of prothrombin time (PT), between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of partial thromboplastin time (PTT) | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of partial thromboplastin time (PTT), between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of bilirubin | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of bilirubin, between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of aspartate aminotransferase (ASAT) | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of aspartate aminotransferase (ASAT), between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of creatinine | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of creatinine, between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of lactate | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of lactate, between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of albumin | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of albumin, between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Time-course of international normalized ratio (INR) | Within the first 7 postoperative days
  Difference in laboratory data, measured by the time-course of international normalized ratio (INR) levels, between the two study arms postoperatively until discharge from ICU or POD 7 (whichever occurs first)
Postoperative peak of blood lactate | During ICU stay, maximum POD 7
  Difference in postoperative peak of blood lactate between the two study groups until discharge from ICU or POD 7 (whichever occurs first)
Length of ICU stay | Until postoperative day 30
  Difference in ICU length of stay between the two study arms
Length of hospital stay | Until postoperative day 30
  Difference in hospital length of stay between the two study arms
Postoperative mortality | Until postoperative day 30
  Difference in mortality between the two study arms until postoperative day 30
Adverse events | Until postoperative day 30
  Difference in quality and quantity of adverse events between the two study arms
Difference in mortality, assessed by 30 days follow up via phone | Postoperative day 30
  Difference in mortality between the two study arms
Difference in coagulation disorder, assessed by 30 days follow up via phone | Postoperative day 30
  Difference in coagulation disorder between the two study arms
Difference in re-admission to hospital, assessed by 30 days follow up via phone | Postoperative day 30
  Difference in re-admission to hospital between the two study arms
Difference in other adverse events, assessed by 30 days follow up via phone | Postoperative day 30
  Difference in other adverse events between the two study arms

CONTACTS AND LOCATIONS:
Overall Officials: Ana Kowark, MD, Principal Investigator — RWTH Aachen University Hospital; Mark Coburn, MD, PhD, Study Director — RWTH Aachen University Hospital
Locations (1):
- University Hospital RWTH Aachen University, Department of Anesthesiology, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No